CLINICAL TRIAL: NCT03754309
Title: A Phase 2a, Randomized, Double Blind, Placebo Controlled, Parallel Group, Multicentre Study of an Anti OX40L Monoclonal Antibody (KY1005) in Moderate to Severe Atopic Dermatitis
Brief Title: A Study of KY1005 in Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kymab Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY1005-CT02; 2018-002299-41 (EudraCT Number); ACT17369 (Other: Sanofi)
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Primary analysis up to day 113. Long term follow up to day 253 (dependent on response).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- KY1005 lower dose (Experimental): Low dose KY1005
  Interventions: Drug: KY1005
- KY1005 higher dose (Experimental): High dose KY1005
  Interventions: Drug: KY1005
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KY1005 — A human anti-OX40 ligand monoclonal antibody
  Other Names: SAR445229
  Arms: KY1005 higher dose; KY1005 lower dose
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
The purpose of this research study is to investigate if KY1005 results in improvement of eczema when given to participants with moderate to severe disease. Side effects of KY1005 will also be explored.

DETAILED DESCRIPTION:
Phase 2a, randomized, double-blinded, placebo-controlled study to evaluate the efficacy, safety and tolerability of two doses of KY1005 in adults with moderate to severe atopic dermatitis whose disease cannot be adequately controlled with topical medications or for whom topical treatment is medically inadvisable.

ELIGIBILITY:
Inclusion Criteria:

* Adults (greater than or equal to [>=] 18 years but less than [<] 75 years of age) with Atopic Dermatitis (AD) for 1 year or longer at Baseline (Day 1; prior to first administration of Investigational Medicinal Product [IMP]).
* Eczema Area and Severity Index (EASI) of 12 or higher at the Screening Visit and 16 or higher at Baseline.
* validated Investigator Global Assessment (vIGA) of 3 or 4 at Baseline.
* AD involvement of 10 percent or more of body surface area at Baseline.
* Documented history, within 6 months prior to Baseline, of either inadequate response to topical treatments or inadvisability of topical treatments.
* Must have applied a stable dose of topical bland emollient (simple moisturizer, no additives [e.g., urea]) at least twice daily for at least 7 consecutive days before Baseline.
* Able and willing to comply with requested study visits/telephone visits and procedures.
* Able and willing to provide punch biopsy of both lesional and non-lesional skin at Baseline.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Recent treatment within specific time windows before the baseline visit for the management of atopic dermatitis such as topical or systemic corticosteroids, biologic or investigational therapies and/or phototherapy.
* Known history of or suspected significant current immunosuppression, including history of invasive opportunistic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration.
* Basal and squamous cell skin cancer in the last 3 years prior to Baseline. Any other malignancies in the last 5 years prior to Baseline (excluding in situ cervical carcinoma).
* Severe concomitant illness that would in the Investigator's opinion inhibit the participant's participation in the study, including for example, but not limited to, renal disease, neurological conditions, heart failure and pulmonary disease.
* Laboratory values at the Screening Visit:
* a. Serum creatinine > 1.6 milligrams per deciliter (mg/dL) (141 micromole per liter [mcmol/L]) in female participants and > 1.9 mg/dL (168 mcmol/L) in male participants;
* b. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 × upper limit of normal (ULN);
* c. Platelet count < 100*10^9/L;
* d. Haemoglobin (Hb): Male < 13.5 g/dL and Female <12 g/dL;
* e. White blood cell count (WBCC) < 3.0*10^9/L;
* f. Absolute neutrophil count < 2.0*10^9/L;
* g. Absolute lymphocyte count < 0.5*10^9/L;
* h. Total bilirubin > ULN.
* Participation in any other clinical study, including non-interventional studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Percentage change in Eczema Area and Severity Index (EASI) | Baseline to day 113
Incidence of treatment-emergent adverse events (TEAEs) | Baseline to day 113

SECONDARY OUTCOMES:
Percentage and absolute change from Baseline in EASI over time | Baseline to day 113
Change in epidermal thickness | Baseline to day 113
Change in keratin 16 staining of skin biopsies | Baseline to day 113
Percentage of patients with at least a 50% reduction in EASI (EASI 50) | Baseline to day 113
Percentage of patients with at least a 75% reduction in EASI (EASI 75) | Baseline to day 113
Percentage of patients with at least a 90% reduction in EASI (EASI 90) | Baseline to day 113
Change in Validated Investigator Global Assessment (vIGA) | Baseline to day 113
Percentage of patients with a response of vIGA 0 or 1 | Baseline to day 113
Change in SCORing of Atopic Dermatis (SCORAD) Index | Baseline to day 113
Change in affected body surface area (BSA) | Baseline to day 113
Change in Patient Orientated Eczema Measure (POEM) | Baseline to Day 113
Change in Patient Orientated SCORing of Atopic Dermatitis (PO-SCORAD) Index | Baseline to day 113
Change in Dermatology Quality of Life Index (DLQI) | Baseline to Day 113
Change in Numerical Rating Scale (NRS) for pruritus | Baseline to day 113

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Weidinger, MaHM, Principal Investigator — University Hospital Schleswig-Holstein, 24105 Kiel, Germany
Locations (19):
- Germany (2):
  - Kymab investigational site 106, Kiel
  - Kymab investigational site 113, Leipzig
- Poland (11):
  - Kymab investigational site 207, Gdansk
  - Kymab investigational site 216, Katowice
  - Kymab investigational site 206, Krakow
  - Kymab investigational site 212, Krakow
  - Kymab investigational site 213, Krakow
  - Kymab investigational site 214, Krakow
  - Kymab investigational site 203, Olsztyn
  - Kymab investigational site 210, Poznan
  - Kymab investigator site 201, Rzeszów
  - Kymab investigational site 204, Warsaw
  - Kymab investigational site 202, Wroclaw
- Spain (4):
  - Kymab investigational site 304, Córdoba
  - Kymab investigational site 303, Madrid
  - Kymab investigational site 302, Seville
  - Kymab investigational site 315, Valencia
- United Kingdom (2):
  - Kymab investigational site 420, Harrogate
  - Kymab investigational site 402, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org